CLINICAL TRIAL: NCT05496413
Title: Investigating the Cognitive Source of Visual Working Memory Impairment in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Wang Jiunn-Kae, Attending psychiatrist, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: N202003153
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Memory Deficits Schizophrenia Neurostimulator; Complications
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active comparator Within group (Experimental): This project will use the StarStim DC stimulator manufactured by Neuroelectrics that was imported with TFDA approval. At the beginning, the participants would be allowed to perform the task which would be followed by application of tACS. The tACS application would be comprised of sham vs active where the sham condition would be given for 30 seconds while the active session would be applied for 15 mins. In tACS, 1mA of theta (6Hz) tACS would be given at the right F4 and P4 electrodes (5*5 cm2, Sponstim® 25). After tACS, the participants would be asked to perform the same task again and the scores (before and after tACS) will be compared and analyzed statistically. Therefore, each patient will need to participate in 2 sessions (active vs. sham), and they will not know which day is which (randomized order).
  Interventions: Device: STARSTIM
- Sham comparator Within group (Sham Comparator): This project will use the StarStim DC stimulator manufactured by Neuroelectrics that was imported with TFDA approval. At the beginning, the participants would be allowed to perform the task which would be followed by application of tACS. The tACS application would be comprised of sham vs active where the sham condition would be given for 30 seconds while the active session would be applied for 15 mins. In tACS, 1mA of theta (6Hz) tACS would be given at the right F4 and P4 electrodes (5*5 cm2, Sponstim® 25). After tACS, the participants would be asked to perform the same task again and the scores (before and after tACS) will be compared and analyzed statistically. Therefore, each patient will need to participate in 2 sessions (active vs. sham), and they will not know which day is which (randomized order).
  Interventions: Device: STARSTIM

INTERVENTIONS:
Device: STARSTIM — In order to evaluate the working memory ability of schizophrenic participants, a task was designed that needs to be performed by them. Firstly, a stimulus of six different color circles of same size in a gray background would be given for 500ms. This would be followed by 2000ms delay phase and then a test array would be appeared. The test array would be exactly same to the stimulus array but with or without change in color of only one circle. The test array would appear on the screen till the participants record their response and they would be asked to respond if the test array matches to the stimulus or not.

SUMMARY:
The investigators plan to investigate the effect of enhancement on visual working memory (VWM) in patients of chronic schizophrenia and determine the predictive factors of effective treatment.

DETAILED DESCRIPTION:
Schizophrenia is a complex neuro-psychiatric disorder that affects a significant portion of total population worldwide. The disease impairs multiple aspects of human cognition, of which visual working memory (VWM) impairment is known to be one of the pivotal cognitive dysfunction in schizophrenic patients. Despite of several attempts that have been made to establish competent treatment strategies to impede cognitive dysfunction of schizophrenia, till date no such studies exhibited satisfactory outcomes. In this context, numbers of studies have been carried out to utilize transcranial direct current stimulation (tDCS) as a treatment option to enhance working memory deficit in various neuropsychiatric populations, but with very limited success. To this end, the present proposal will focus on the use of transcranial alternating current stimulation (tACS) to better target the oscillatory mechanisms underlying VWM. Our specific aims are twofold, namely, 1) Does DLPFC tACS work on schizophrenic patients in terms of VWM improvement, and 2) how is tACS facilitating patients' VWM? This is because VWM deficit can be caused by poor encoding, poor maintenance, or poor retrieval (or any combination between them). Failure at any of those steps will make the patients appear to have poor VWM from clinical observation, but the cognitive process that is impaired may not be the same across populations.

ELIGIBILITY:
Inclusion Criteria:

1. Inform consent acquired
2. Age 20 to 65
3. Right-handed
4. Patients with schizophrenia diagnosed according to DSM-5 criteria

Exclusion Criteria:

1. Participants who are pregnant or breastfeeding
2. Participants who have metal implants
3. Participants who have alcohol/substance use disorder or received electro-convulsive therapy within the past 6 months.
4. Participants who have history of head injury with loss of consciousness
5. Participants who have history of brain lesions, infection, or epilepsy
6. Skin lesions on the electrodes placed
7. Cancer patients
8. Patients with high fever
9. Patients with significant sensory loss

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
VWM dysfunction | up to one hour
  Using the VWM task, investigate at which time point (encoding stage, maintenance stage, or retrieval stage) is VWM dysfunction occurring in schizophrenia patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jiunn-Kae Wang, MD, MSc, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No